CLINICAL TRIAL: NCT00469833
Title: Pathogenesis of the Impaired Incretin Effect in Type 2 Diabetes
Brief Title: Insulin Secretion in Diabetes Before and After Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDA-010-06S
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Hyperglycemia
Keywords: Diabetes; Glucose Tolerance; Incretin; Insulin
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Insulin Resistance | interventions — Insulin Glargine; Insulin, Long-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Intervention: Insulin glargine treatment. The study is designed as a within subjects comparison of insulin secretion in type 2 diabetic patients before and after 2 months of insulin treatment to reduce blood glucose. Insulin secretion will be determined with a hyperglycemic clamp using 20% dextrose, and ingestion of an oral glucose solution (75 g).
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin glargine — Diabetic subjects will be treated with insulin glargine once daily for 2 months. Subjects will monitor their blood glucose and have their insulin dose adjusted in steps of 4-6 units to achieve a goal of less than or equal to 120 mg/dl for fasting blood glucose.
  Other Names: Basal insulin; Long-acting insulin; Lantus

SUMMARY:
The objective of this project is to understand defects in insulin secretion that contribute to abnormal glucose metabolism in patients with diabetes. In particular the effects of signals released from the intestine to stimulate insulin secretion will be tested. Patients with type 2 diabetes will have insulin secretion in response to glucose and intestinal factors before and after insulin treatment to lower their blood glucose. It is expected that the results of this work will provide valuable information for treating diabetic people.

DETAILED DESCRIPTION:
The objective of this project is to understand defects in insulin secretion that contribute to abnormal glucose metabolism in patients with diabetes. Diabetes is a major problem for patients receiving care at VA medical centers among whom 20% are affected. Specifically, this project will seek to determine the mechanism(s) by which the incretin effect is impaired in diabetic patients. The incretin effect refers to the action of GI hormones and neural stimuli to increase insulin secretion after food intake, and accounts for approximately 50% of postprandial insulin secretion in nondiabetic humans. There are several studies indicating that this response is severely impaired in patients with type 2 diabetes. The mechanism(s) by which this occurs has not been explained. There is some evidence to suggest that secretion of the important incretins, glucagon-like peptide 1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP), may be impaired in diabetic individuals. There is also some data to suggest that the beta-cells in persons with diabetes are insensitive to the incretins. The problem with the current state of knowledge in this area is that previous work has involved small numbers of diabetic subjects, and did not directly test mechanisms by which the incretin effect is altered in diabetes.

In this project we will determine the role of hyperglycemia to impair the incretin effect. Type 2 diabetic subjects will have the incretin effect measured before and after intensified diabetes treatment. This study will test the effect of chronic hyperglycemia on incretin mediated insulin secretion. In all studies, the incretin effect will be measured before and after these interventions using studies with a within subjects design. A combined glucose clamp/meal tolerance test protocol will be used to quantify the incretin effect.

These studies will allow the role of incretin secretion, incretin action, and overall metabolic milieu, on postprandial insulin secretion to be defined. The results of these studies will add important new information for understanding abnormal beta-cell function in diabetes. By identifying the sites where the incretin effect is impaired this project will provide the basis for new approaches to treat diabetic patients. This is especially relevant with the recent availability of new medications that target the incretin pathways to lower blood glucose.

The blood samples will be drawn and processed in the GCRC. The samples will be frozen and stored in Building 15, Room 401. Samples will be shipped to the Genome Research Institute by staff trained in IATA shipping procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1:

  * (non-diabetics)

    * male/female 30-65 yrs old,
    * free of active medical disease,
    * no history of diabetes.
  * (diabetics)

    * HbA1c=6.5-8.5,
    * treated with metformin, a sulfonylurea, or combination,
    * Stable body wt with BMI 28-40.
* Aim 2: Same as above
* Aim 3: Diabetic with HgA1c 8.0-9.5

Exclusion Criteria:

* Aim 1: For both groups: no history of: pancreatitis, cardiac, gastrointestinal, renal or liver disease.
* Aim 2: Same as above
* Aim 3: Same as above, plus a diagnosis of incipient diabetic nephropathy severe nonproliferative, or proliferative retinopathy.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — Cincinnati VA Medical Center
Locations (1):
- VA Medical Center, Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Result] An Z, Prigeon RL, D'Alessio DA. Improved glycemic control enhances the incretin effect in patients with type 2 diabetes. J Clin Endocrinol Metab. 2013 Dec;98(12):4702-8. doi: 10.1210/jc.2013-1199. Epub 2013 Oct 3. PMID 24092826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from VAMC from 2010-2012
Pre-assignment Details: No subjects excluded
Groups:
- Uncontrolled Type 2 Diabetic Subjects: Eligible subjects will have measures of insulin secretion measured using the OGTT/hyperglycemic clamp technique before and after 2 months of treatment to lower blood glucose.
Period: Overall Study
Arm/Group | Uncontrolled Type 2 Diabetic Subjects
Started | 17 (17 subjects met inclusion criteria and consented for the study)
Completed | 15
Not Completed | 2
Not completed — No IV access | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Within subjects comparison; before and after treatment.
  Beta-cell function measured with OGTT/hyperglycemic clamp
Arm/Group | Arm 1
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: ISR in Response to a Glucose Clamp and Oral Glucose Ingestion Before and After 2 Months of Insulin Treatment to Improve Average Glycemia.
Description: Subjects had glucose clamps for 270 minutes with serial sampling of blood for measurement of insulin and C-peptide. At 90 minutes into the clamp they consumed 75 g of oral glucose solution. Meal-stimulated insulin secretion was summarized as the mean plasma C-peptide from 90-270 minutes. This outcome measure was compared for each subject before treatment and after 2 months of insulin treatment to lower blood glucose. Subjects were started on 20 units of insulin glargine after their first visit and asked to measure their morning blood glucose daily. The dose of insulin was increased in increments of 4-6 units every 3 days targeting an average morning glucose level of less then 120 mg/dl. After 2 months of treatment the primary outcome was repeated with a second glucose clamp / oral glucose tolerance test, identical to the first.
Time Frame: 180 minutes
Measure: Mean (Standard Error); unit: pmol/min
Groups:
- Oral Glucose: Oral glucose administered to uncontrolled type 2 diabetic subjects.
- IV Glucose: IV glucose administered to uncontrolled type 2 diabetic subjects.
Arm/Group | Oral Glucose | IV Glucose
Number analyzed (Participants) | 15 | 15
pmol/min
  Insulin secretion at baseline | 0.67 (0.07) | 0.75 (0.10)
  Insulin secretion at 8 weeks | 1.11 (0.22) | 0.76 (0.11)

2. Primary Outcome: C-peptide Concentration in Response to a Glucose Clamp and Oral Glucose Ingestion Before and After 2 Months of Insulin Treatment to Improve Average Glycemia.
Description: as for outcome 1
Time Frame: 180 minutes
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Oral Glucose | IV Glucose
Number analyzed (Participants) | 15 | 15
nmol/L
  C-peptide at baseline | 7.10 (0.92) | 5.63 (0.97)
  C-peptide at 8 weeks | 10.89 (2.20) | 6.02 (0.88)

3. Primary Outcome: Insulin Concentration in Response to a Glucose Clamp and Oral Glucose Ingestion Before and After 2 Months of Insulin Treatment to Improve Average Glycemia.
Description: as for outcome 1
Time Frame: 180 minutes
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Oral Glucose | IV Glucose
Number analyzed (Participants) | 15 | 15
pmol/L
  Insulin at baseline | 546.9 (162.6) | 316.4 (59.0)
  Insulin at 8 weeks | 934.6 (282.2) | 395.6 (106.3)

4. Secondary Outcome: HbA1c Before and After 2 Months of Insulin Treatment to Improve Average Glycemia.
Description: Type 2 diabetic subjects had HbA1c measured before and after 2 months of basal insulin glargine treatment.
Time Frame: 2 months
Measure: Mean (Standard Error); unit: % glycosylated hemoglobin
Arm/Group | Uncontrolled Type 2 Diabetic Subjects
Number analyzed (Participants) | 15
% glycosylated hemoglobin
  HbA1c at baseline | 8.6 (0.2)
  HbA1c at 8 weeks | 7.1 (0.2)

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Two subjects could not complete the initial assessment due to poor IV access. All 15 subjects who completed the initial assessment and were started on insulin completed the study. There were no significant adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No